CLINICAL TRIAL: NCT00943696
Title: Effects of White Wine vs. Tea Intake During and an Alcoholic Digestive Following a High Fat, High Calorie Cheese Fondue Meal on Gastric Emptying and Abdominal Symptoms in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: COOP (Unknown)
Responsible Party: Dr. Mark Fox, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Fonduestudie_EKGs
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Ingestion of white wine vs. tea during and an alco — 4 x 50ml glasses of white wine (12% alcohol) or tea will be taken according to a randomization scheme After the meal 1 x 20ml of Kirsch (40% alcohol) or tea will be taken

SUMMARY:
Tradition holds that the intake of different drinks with a meal has an important influence on the digestion of food and postprandial symptoms such as fullness, bloating and satiety; however this assumption have never been subjected to controlled study

A classic example is the Swiss cheese fondue. The intake of white wine, tea and cherry schnapps (Kirsch) are often attributed either positive or negative effects on the gastrointestinal tract.

In this study the effect of white wine vs. tea intake during and an alcoholic digestive following a high fat, high calorie Swiss fondue meal on gastric emptying and visceral perception will be investigated using a randomized, controlled study design.

The fondue will be labeled with non-radioactive 13C octanoate for assessment of gastric emptying by breath-test.

ELIGIBILITY:
Inclusion criteria: • able to communicate well with the investigators and provide written consent

• Body Mass Index: 19-30 kg/m2

Exclusion criteria: • physical co-morbidity requiring active treatment

* psychiatric (DSM IV) disorders limiting the ability to comply with study
* use of medications influencing upper GI motility
* evidence of current drug or alcohol abuse
* history of gastrointestinal disease or surgery except appendicectomy or hernia repair

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Effect of white wine vs. tea on gastric emptying | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Heinrich H, Goetze O, Menne D, Iten PX, Fruehauf H, Vavricka SR, Schwizer W, Fried M, Fox M. Effect on gastric function and symptoms of drinking wine, black tea, or schnapps with a Swiss cheese fondue: randomised controlled crossover trial. BMJ. 2010 Dec 14;341:c6731. doi: 10.1136/bmj.c6731. PMID 21156747